CLINICAL TRIAL: NCT06889727
Title: Pregnancy and Childbirth in Women with Thalassemia Yesterday and Today: a Multicentre Observational Study
Brief Title: Pregnancy and Childbirth in Women with Thalassemia Yesterday and Today
Status: Completed | Type: Observational
Sponsor: Fondazione per la Ricerca sulle Anemie ed Emoglobinopatie in Italia (Other)
Responsible Party: Sponsor
Other Study IDs: GRAV001
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Thalassemia
MeSH Terms: conditions — Thalassemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Recent advances in the management of thalassemia have significantly improved life expectancy and quality of life of patients with this hemoglobinopathy, with a consequent increase in their reproductive potential and desire to have children.Since an initial report of a successful pregnancy in a woman with thalassemia major by Walker in 1969, hundreds of pregnancies have been reported so far, highlighting that women carefully managed in the preconception phase usually carry out a successful gestation and labor, both in case of spontaneous conception and assisted reproductive techniques.

ELIGIBILITY:
Inclusion Criteria:

* Transfusion dependent and nontransfusion- dependent thalassemia
* Pregnancy ended with the birth of a live or dead foetus
* Pregnancy ended in miscarriage or voluntary abortion
* Pregnancy in progress

Exclusion Criteria:

* Other types of anemia
* Pregnancy not initiated despite assisted fertilization practices
* Subjects unwilling to sign informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — FEMALE
Study Population: FEMALE THALASSEMIE DEPEND TRANSFUSION
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2023-08-09 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-05-14 (Actual)

PRIMARY OUTCOMES:
number of pregnancies in women with beta thalassemia followed in Italian centres | 15 YEARS
  To evaluate the number of pregnancies in women with beta thalassemia followed in Italian centres and how the increase in the average age of the thalassemia population impact on the number of new pregnancies over time
number of pregnancies spontaneously | 15 YEARS
  many pregnancies occurred spontaneously
number of pregnancies after hormonal stimulation | 15 YEARS
  number of pregnancies after hormonal stimulation
likelihood of miscarriage | 15 YEARS
  To evaluate the likelihood of miscarriage
foetal death | 15 YEARS
  To evaluate foetal death

CONTACTS AND LOCATIONS:
Locations (1):
- UniversityCagliari, OspPed Microcitemico, Cagliari, Cagliari, CAGLIARI, Italy

IPD SHARING:
Plan to Share IPD: No